CLINICAL TRIAL: NCT00740532
Title: Observational Study Assessing Molecular Features Predicting Response/Resistance to Trastuzumab in Metastatic Breast Cancer Patients
Brief Title: Molecular Features Predicting Response/Resistance to Trastuzumab in Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Armando Santoro, MD, Istituto Clinico Humanitas
Other Study IDs: ONC/OSS-01/2007
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Breast Cancer
Keywords: EGFR, HER-2, HER-3, MET, KRAS
MeSH Terms: conditions — Breast Neoplasms; Lethal Congenital Contracture Syndrome 2 | interventions — In Situ Hybridization, Fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paraffine embedded tumor sections
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Breast cancer patients treated with Herceptin-based therapy
  Interventions: Genetic: Gene mutation analyses and FISH

INTERVENTIONS:
Genetic: Gene mutation analyses and FISH — FISH and mutation analyses of multiple genes

SUMMARY:
Aim of the study is to assess the impact on response to Herceptin-based therapy in patients with advanced breast cancer. Tumor specimens from primary breast cancer will be analized for several biological factors potentially involved in Herceptin sensitivity.

Tests that will be performed include: FISH analyses of EGFR, HER-2, HER-3, C-MYC, PTEN, MET, IGFR-1. Immunofluorecence of P95HER2. Mutation analyses of EGFR, HER-2, MET, C-MYC, PTEN, KRAS, PIK3CA, IGFR-1. Immunohistochemistry of the same biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Hystological diagnosis of breast cancer
* Availability of tumor tissue
* Availability to assess the response to Trastuzumab according to RECIST criteria
* Availability of clinical data

Exclusion Criteria:

* Unavailability of tumor tissue
* Impossibility to assess the response to Trastuzumab according to RECIST criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients treated with Herceptin-based therapy
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Association of a specific biomarker with response to Herceptin-based therapy | Response after two months of treatment

SECONDARY OUTCOMES:
Association of a specific biomarker with time to progression survival and patient's characteristics | At the end of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy